CLINICAL TRIAL: NCT07310849
Title: Digital Care Community Common Good Program Enhances Holistic Health Management for Middle Aged and Older Adults With Diabetes Mellitus and Multiple Chronic Conditions
Brief Title: Digital Care for Holistic Health in Older Adults With Diabetes and Multimorbidity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB 24 021 B1
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Type2Diabetes; Hypertension; Dyslipidemia; CKD; Cardio Vascular Disease; Gout Arthritis
Keywords: community care; diabetes mellitus; multimorbidity; quality of life; self-management
MeSH Terms: conditions — Hypertension; Dyslipidemias; Arthritis, Gouty; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group receives usual care and a 6-month Digital Care Community Common Good program (Experimental): online and in-person educational sessions, telephone care, use of the mHealth platform (featuring educational, data monitoring, contextual learning, interactive, and reminders), as well as home visits, case discussions, and individualized care plans for high-risk cases.
  Interventions: Behavioral: Digital Care Community Common Good Program
- The control group that receives usual care and the local integrated medical network information (Other): receives usual care and the local integrated medical network information, including clinics and healthcare institutes that provide comorbidity care and counseling.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Digital Care Community Common Good Program — a 6-month Digital Care Community Common Good program (online and in-person educational sessions, telephone care, use of the mHealth platform (featuring educational, data monitoring, contextual learning, interactive, and reminders), as well as home visits, case discussions, and individualized care plans for high-risk cases.)
  Arms: The experimental group receives usual care and a 6-month Digital Care Community Common Good program
Behavioral: Usual Care — receives usual care and the local integrated medical network information, including clinics and healthcare institutes that provide comorbidity care and counseling.
  Arms: The control group that receives usual care and the local integrated medical network information

SUMMARY:
The purpose of this study was to explore the effectiveness of the "Digital Care Community Common Good" program in improving disease control indicators, self-management abilities, depression, and quality of life among patients with comorbidities and type 2 diabetes. The study was designed as a two-year experimental study, with a specific area in New Taipei City selected as the research site. In the first year, the main tasks include establishing an integrated intervention team composed of primary healthcare providers and community resources, expanding the functionalities of the mHealth platform, developing digital educational materials for diabetes comorbidities care, and recruiting and training 6 to 8 community care volunteers. Additionally, 169 eligible participants with type 2 diabetes and comorbidities will be recruited from four communities, completing baseline assessments and randomization into groups. In the second year, a 6-month intervention and effectiveness evaluation of the " Digital Care Community Common Good " program will be implemented. The intervention includes online and in-person educational sessions, telephone care, use of the mHealth platform (featuring educational, data monitoring, contextual learning, interactive, and reminders), as well as home visits, case discussions, and individualized care plans for high-risk cases. Disease control indicators, selfmanagement abilities, depression, and quality of life will be tracked immediately post-intervention, at 3 month, and at 6 month to assess outcomes and changes over time. This study expects to enhance health management for diabetes patients with comorbidities through digital care and interdisciplinary collaboration, offering evidence-based insights and recommendations for policy implementation in the integration of community and primary healthcare models.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Consent: Individuals aged 50 years or older who are willing to provide written informed consent.
2. Language and Literacy: Participants must be literate and able to communicate in Mandarin or Taiwanese.
3. Medical Diagnosis: Participants must have a physician-confirmed diagnosis of type 2 diabetes mellitus (T2DM) and at least one comorbid chronic disease (e.g., hypertension, hyperlipidemia, chronic kidney disease, or heart disease).
4. Technology Use: Participants must own a smartphone and be willing to use the LINE messaging app and web-based health education links.
5. Residence: Participants must reside within one of the four participating communities and have no plans to move away during the study intervention period.

Exclusion Criteria:

* (1)Those with severe diabetes-related complications, such as renal failure, cerebrovascular disease, diabetic foot, or retinopathy.

  (2)Individuals with psychiatric disorders, undergoing active cancer treatment, or those unable to perform independent self-care (e.g., due to visual impairment or mobility limitations).

  (3)Individuals without diabetes but with other chronic diseases. (4)Individuals residing in long-term care institutions. (5)Individuals who are simultaneously participating in other intervention programs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The Disease Self-Management Scale | T0 Pre-Test: Conducted before the intervention. T1: Conducted immediately after completing the intervention. T2: Conducted three months after completing the intervention. T3: Conducted six months after completing the intervention.
  This study employs the Disease Self-Management Scale by Professor Ching-Min Chen (2012), based on the Chronic Disease Care Management Model.
  The scale includes 39 items across four subscales: Partnership, Self-care performance, Problem-solving, and Emotional management. Each item is rated on a 4-point Likert scale (0-3), reflecting participants' self-management behaviors over the past three months. Higher scores indicate better self-management ability. The scale has been validated in community-based studies involving older adults with multiple metabolic chronic diseases, demonstrating strong reliability and validity. Cronbach's alpha (total scale): .83. Subscales: Partnership (.88), Self-care activities (.78), Problem-solving (.90), Emotional management (.60). Internal consistency is considered satisfactory.

CONTACTS AND LOCATIONS:
Locations (1):
- Wugu District Public Health Center,, New Taipei City, Wugu District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dattani I, Ganatra S. Oral manifestations of HIV infections. Oral Health. 1993 Jul;83(7):15-7. No abstract available. PMID 8272348
- [Background] Bredell F. Wait! What's not trash--it's recyclable! Mich Hosp. 1991 May;27(5):26-30. No abstract available. PMID 10110949
- [Background] Espeland MA, Gaussoin SA, Bahnson J, Vaughan EM, Knowler WC, Simpson FR, Hazuda HP, Johnson KC, Munshi MN, Coday M, Pi-Sunyer X. Impact of an 8-Year Intensive Lifestyle Intervention on an Index of Multimorbidity. J Am Geriatr Soc. 2020 Oct;68(10):2249-2256. doi: 10.1111/jgs.16672. Epub 2020 Jul 17. PMID 33267558
- [Background] Davis J, Fischl AH, Beck J, Browning L, Carter A, Condon JE, Dennison M, Francis T, Hughes PJ, Jaime S, Lau KHK, McArthur T, McAvoy K, Magee M, Newby O, Ponder SW, Quraishi U, Rawlings K, Socke J, Stancil M, Uelmen S, Villalobos S. 2022 National Standards for Diabetes Self-Management Education and Support. Diabetes Care. 2022 Feb 1;45(2):484-494. doi: 10.2337/dc21-2396. No abstract available. PMID 35050365
- See also: Available upon reasonable request from the Principal Investigator. — https://webmis.cgust.edu.tw/Research/T_View.asp?TSn=53